CLINICAL TRIAL: NCT05007626
Title: Association of Axial Length and Refraction With Near Horizontal Heterophoria in Chinese Children
Brief Title: Near Horizontal Heterophoria in Chinese Children
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Principal Investigator, Yan Wang, Director, Head of Ophthalmology, Tianjin Eye Hospital
Other Study IDs: 2021020
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- zero to six Exo
  Interventions: Other: axial length and refractive error

INTERVENTIONS:
Other: axial length and refractive error — Comparing the correlation between heterophoria and refraction, even after age adjustment.

SUMMARY:
This study aimed to assess the association of refraction and axial length with near-horizontal heterophoria in a large population-based study of school-aged Chinese children. The study makes a significant contribution to better know the etiology of myopia progression and ocular axial length development. Further, this study will be of interest to the readership of your journal because its noteworthy finding and which could contribute to guide recommendations for targeted interventions to slow myopia progression.

DETAILED DESCRIPTION:
Myopia is becoming a global public health burden which is believed to have a multifactorial etiology. The relationship between heterophoria and refraction remains controversial. We describe the association of refraction and axial length (AL) with heterophoria in a large population-based study of school-aged Chinese children. Eleven thousand thirteen elementary school children grades 1-6, were included in this school-based, cross-sectional study. Near phoria data was quantified by using Maddox rod test and prism at 33 cm. Children in each grade level were sorted into three groups based upon phoria: 1) those with more than six prism diopters (PD) exophoria, 2) those with zero to six PD exophoria, and 3) those with any amount of esophoria. Autorefraction was measured by autorefractor (Topcon KR8900, Japan) and AL was measured by Optical Biometer AL-Scan (Nidek AL-Scan, Japan). A generalized additive model (GAM) was applied with a Gaussian link to explore the association between the refractive error or axial length and heterophoria. An additional age-adjusted model was also employed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* ages of 6 and 13 years
* Chinese school children

Exclusion Criteria:

* Subjects with eye diseases or strabismus

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 15,081 Chinese children between the ages of 6 and 13 years were enrolled in this study. Subjects with eye diseases or strabismus were excluded, so data validated from 11,013 children were used for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 15081 (Actual)
Dates: Start 2017-01-29 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
refractive error | change from baseline with EDTRS chart at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

REFERENCES:
- [Background] Grzybowski A, Kanclerz P, Tsubota K, Lanca C, Saw SM. A review on the epidemiology of myopia in school children worldwide. BMC Ophthalmol. 2020 Jan 14;20(1):27. doi: 10.1186/s12886-019-1220-0. PMID 31937276
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007